CLINICAL TRIAL: NCT01614756
Title: A Two-Part, Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Dose, Dose-Escalation Study of Subcutaneous and Intravenous Administration of IL-31 mAb (Anti-Interleukin 31 Monoclonal Antibody; BMS-981164) in Healthy Subjects and Adult Subjects With Atopic Dermatitis
Brief Title: A Two-Part, Phase 1, Single-Dose Study of IL-31 mAb (Anti-Interleukin 31 Monoclonal Antibody); in Healthy Subjects and Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM134-002; 2012-001865-34 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Subjects and Atopic Dermatitis Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- Dose Escalation-BMS-981164 (0.1 mg/kg) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 0.1 mg/kg solution subcutaneously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution subcutaneously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (0.01 mg/kg) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 0.01 mg/kg solution subcutaneously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution subcutaneously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (0.03 mg/kg) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 0.03 mg/kg solution subcutaneously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution subcutaneously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (0.06 mg/kg) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 0.06 mg/kg solution subcutaneously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution subcutaneously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation- BMS-981164 (0.1 mg/kg) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 0.1 mg/kg solution subcutaneously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution subcutaneously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (0.3 mg/kg) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 0.3 mg/kg solution subcutaneously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution subcutaneously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (1 mg/kg SC) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 1 mg/kg solution subcutaneously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution subcutaneously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (1 mg/kg IV) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 1 mg/kg solution intravenously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution intravenously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (3 mg/kg IV) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 3 mg/kg solution intravenously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution intravenously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation-BMS-981164 (10 mg/kg IV) or Placebo (Experimental): Part 1
  Single dose of BMS-981164 10.0 mg/kg solution intravenously
  OR
  Single dose of Placebo matching with BMS-981164 0 mg/kg solution intravenously
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation- BMS-981164 or Placebo (dose group 1) (Experimental): Part 2
  BMS-981164: Solution, Depending on dose level selected could be subcutaneous or IV, 3 mg/kg, once, single dose
  OR
  Placebo matching with BMS-981164: Solution, Depending on dose level selected could be subcutaneous or IV, 0 mg, once, single dose
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation- BMS-981164 or Placebo (dose group 2) (Experimental): Part 2
  BMS-981164: Solution, Depending on dose level selected could be subcutaneous, 0.1 mg/kg, once, single dose
  OR
  Placebo matching with BMS-981164: Solution, Depending on dose level selected could be subcutaneous, 0 mg, once, single dose
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation- BMS-981164 or Placebo (dose group 3) (Experimental): Part 2
  BMS-981164: Solution, Depending on dose level selected could be subcutaneous, ≤ 0.1 mg/kg, once, single dose
  OR
  Placebo matching with BMS-981164: Solution, Depending on dose level selected could be subcutaneous, 0 mg, once, single dose
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164
- Dose Escalation- BMS-981164 or Placebo (dose group 4) (Experimental): Part 2
  BMS-981164: Solution, Depending on dose level selected could be subcutaneous, ≤ 3.0 mg/kg and >1.0mg/kg, once, single dose
  OR
  Placebo matching with BMS-981164: Solution, Depending on dose level selected could be subcutaneous, 0 mg, once, single dose
  Interventions: Biological: BMS-981164; Biological: Placebo matching with BMS-981164

INTERVENTIONS:
Biological: BMS-981164
  Other Names: IL-31 mAB
Biological: Placebo matching with BMS-981164

SUMMARY:
The purpose of the study is to determine safety and tolerability of IL-31 mAB

DETAILED DESCRIPTION:
Healthy Volunteers not acceptable for "Part 2" (Adult subjects with Atopic Dermatitis)

Enrollment: (both Part 1 and Part 2) Part 2 will consist of up to 42 patients with atopic dermatitis

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Part 1: Healthy subjects
* Part 2: Adult subjects with:

  1. Atopic dermatitis severity as assessed by Physician Global Assessment rating of 3 or higher (i.e., moderate or greater) on a scale of 0 to 5
  2. Pruritus severity of at least 7 of 10 on a visual analog scale

Exclusion Criteria:

* Receipt of systemic immunosuppressants, other than biological agents, or topical calcineurin inhibitors (tacrolimus or pimecrolimus) within 4 weeks prior to study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
For both Part 1 and Part 2, the primary endpoint will be based on incident adverse event reports, vital sign measurements, physical (including injection site) examinations, electrocardiograms (ECGs), medical history, and clinical laboratory tests | Up to 16 weeks after single dose

SECONDARY OUTCOMES:
The Maximum observed serum concentration (Cmax) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Time of maximum observed serum concentration (Tmax) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Area under the serum concentration-time curve from zero to time of the last quantifiable concentration [AUC(0-T)] of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Terminal serum half-life (T-HALF) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Apparent volume of distribution at steady state (Vss/F) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Volume of distribution at steady state (Vss) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Apparent total body clearance (CLT/F) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Total body clearance (CLT) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
The Absolute bioavailability (F) of BMS-981164 will be derived from serum concentration versus time | 13 timepoints upto 16 weeks after single dose
Frequency of subjects with one or more positive post-treatment anti-drug antibodies (ADA) assessments | Up to 16 weeks after single dose
  The Immunogenicity of BMS-981164 will be assessed by this ADA assessments

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United Kingdom (4):
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Newcastle upon Tyne, Tyne and Wear
  - Local Institution, Manchester
  - Local Institution, Nottingham

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx